CLINICAL TRIAL: NCT05543083
Title: Cognitive-Behavioral Therapy and Exercise Training in Adolescents At-Risk for Type 2 Diabetes
Acronym: CBTeX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22-0180; 1R01DK132557-01 (NIH)
Record Dates: First submitted 2022-08-24; First posted 2022-09-16 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Insulin Resistance; Depression; Depressive Disorder; Mood Disorders; Mental Disorder in Adolescence; Hyperinsulinism; Glucose Metabolism Disorders; Metabolic Disease
Keywords: Adolescent Type 2 Diabetes Prevention; Exercise Training
MeSH Terms: conditions — Insulin Resistance; Depression; Depressive Disorder; Mood Disorders; Hyperinsulinism; Glucose Metabolism Disorders; Metabolic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive-Behavioral Therapy followed by Exercise Training (Experimental): 6-week cognitive-behavioral therapy intervention of 6 weekly 1-hour group sessions followed by a 6-week exercise training intervention of 6 weekly 1-hour group sessions
  Interventions: Behavioral: Cognitive-Behavioral Therapy followed by Exercise Training
- Exercise Training followed by Cognitive-Behavioral Therapy (Active Comparator): 6-week exercise training intervention of 6 weekly 1-hour group sessions followed by a 6-week cognitive-behavioral therapy intervention of 6 weekly 1-hour group sessions
  Interventions: Behavioral: Exercise Training followed by Cognitive-Behavioral Therapy
- Exercise Training Only (Active Comparator): 6-week exercise training intervention of 6 weekly 1-hour group sessions followed by an additional 6-week exercise training intervention of 6 weekly 1-hour group sessions
  Interventions: Behavioral: Cognitive-Behavioral Therapy Only
- Cognitive-Behavioral Therapy Only (Active Comparator): 6-week cognitive-behavioral therapy intervention of 6 weekly 1-hour group sessions followed by an additional 6-week cognitive-behavioral therapy intervention of 6 weekly 1-hour group sessions
  Interventions: Behavioral: Exercise Training Only

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy followed by Exercise Training — 6-week group CBT (cognitive-behavioral therapy; 1 hour/week for 6 weeks) followed by 6-week group exercise training (1 hour/week for 6 weeks). Home practice is assigned throughout the 12-week intervention period.
  Other Names: CBT->Exercise Training
  Arms: Cognitive-Behavioral Therapy followed by Exercise Training
Behavioral: Exercise Training followed by Cognitive-Behavioral Therapy — 6-week group exercise training (1 hour/week for 6 weeks) followed by 6-week group CBT (1 hour/week for 6 weeks). Home practice is assigned throughout the 12-week intervention period.
  Other Names: Exercise Training -> CBT
  Arms: Exercise Training followed by Cognitive-Behavioral Therapy
Behavioral: Cognitive-Behavioral Therapy Only — 6-week group CBT (1 hour/week for 6 weeks), with continuation of group CBT for a second 6-week period (1 hour/week for 6 weeks). Home practice is assigned throughout the 12-week intervention period.
  Other Names: CBT Only
  Arms: Exercise Training Only
Behavioral: Exercise Training Only — 6-week group exercise training (1 hour/week for 6 weeks), with continuation of group exercise for a second 6-week period (1 hour/week for 6 weeks). Home practice is assigned throughout the 12-week intervention period.
  Arms: Cognitive-Behavioral Therapy Only

SUMMARY:
The investigators are doing this study to learn more about how to prevent type 2 diabetes in teenage girls. The purpose of this study is to find out if taking part in a cognitive-behavioral therapy group, exercise training group, or a combination of cognitive-behavioral therapy and exercise training groups, decreases stress, improves mood, increases physical activity and physical fitness, and decreases insulin resistance among teenagers at risk for diabetes.

DETAILED DESCRIPTION:
There has been rapid escalation in adolescent-onset type 2 diabetes (T2D), particularly in females from historically disadvantaged racial/ethnic groups. Prevention is critical because adolescent-onset T2D often shows a more aggressive disease course than adult-onset, and effective treatment options remain elusive. Standard-of-care for T2D prevention includes exercise training to ameliorate insulin resistance, a key physiological precursor to T2D. Despite short-term benefits, exercise training shows insufficient effectiveness in adolescents at-risk for T2D. Depression may be explanatory in a considerable subset of teenagers. Adolescence is notable for increases in depression and decreases in physical activity, especially in females with obesity. Youths' depression symptoms contribute to worsening insulin resistance over time, independent of BMI (kg/m2), likely through stress-mediated pathways such as reduced physical activity and fitness. Also, adolescent depression is associated with decreased physical activity and cardiorespiratory fitness, even after accounting for adiposity, and depression predicts greater non-adherence to exercise training. The central theme of this proposal is that an intervention sequence of delivering cognitive-behavioral therapy (CBT) first, followed by intervening with exercise training second, will offer a targeted, efficacious strategy for improving insulin resistance and consequently, lowering T2D risk in adolescent females at-risk for T2D with depression symptoms. In a prior National Institute of Health (NIH) /National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) K99/R00 randomized controlled trial (RCT), the investigators found that 6-week group CBT decreased depression at 6-week follow-up in adolescent females at-risk for T2D with moderately elevated depression, compared to a 6-week didactic health education control group. Adolescents with elevated depression who were randomized to CBT had lower fasting and 2-hour insulin at 1-year vs. controls. Our preliminary data suggest that CBT's focus on enhancing frequency/enjoyment of physical activity to combat depressed mood partially explained why decreasing depression lowered T2D risk. It is not known if CBT is just as efficacious as standard-of-care exercise training, or whether CBT followed by exercise training results in a maximally potent alleviation of T2D risk in adolescent females at-risk for T2D with depression symptoms. To address these gaps and directly build on our prior work, the investigators propose a four-arm RCT to: (1) Compare the efficacy of four 6-week-->6-week sequences for improving insulin resistance in N=300 adolescent females at-risk for T2D with elevated depression symptoms: (i) CBT-->exercise, (ii) exercise-->CBT, (iii) CBT only (CBT-->continue CBT), and (iv) exercise only (exercise-->continue exercise); (2) Evaluate physical activity/fitness as mediators underlying the depression-insulin resistance association; and (3) Evaluate underlying mechanisms by which decreasing depression increases physical activity and improves fitness and insulin resistance using a mixed-methods process evaluation. Findings will support our long-term goal to identify feasible, cost-effective intervention strategies with high potential for effective dissemination to adolescents at-risk for T2D with elevated depression symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 12-17 years
* Body Mass Index (BMI)>= 85 for age and sex
* Type 2 Diabetes (T2D) first-or second-degree relative
* Center for Epidemiologic Studies Depression Scale (CES-D) total score >=21

Exclusion Criteria:

* T2D/ Type 1 Diabetes (T1D) or any major medical condition (e.g. cardiovascular, renal) that would prohibit the ability to participate in exercise training
* Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) conduct disorder, substance abuse/ dependence, obsessive compulsive disorder, panic attacks, post-traumatic stress disorder, anorexia/bulimia, & schizophrenia
* Insulin sensitizers, weight loss medications & chronic steroids
* Structured weight loss treatment or bariatric surgery
* Pregnancy, nursing

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Insulin Resistance | 1-year
  Homeostatic model assessment of insulin resistance (HOMA-IR) estimated from fasting insulin and glucose as part of oral glucose tolerance testing

SECONDARY OUTCOMES:
Insulin sensitivity | 1-year
  Insulin sensitivity index (ISI) derived from fasting and two-hour insulin and glucose as part of oral glucose tolerance testing
Cardiorespiratory fitness | 1-year
  Maximum volume of oxygen (VO2 peak) during cycle ergometry testing using a graded protocol to exertion
Rate Perceived Exertion | 1-year
  Adolescent report on the Borg Scale during cycle ergometry testing
Exercise enjoyment | 1-year
  Adolescent report on the Physical Activity Enjoyment Scale (PACES), total score
Exercise self-efficacy | 1-year
  Adolescent report on the Exercise Self-Confidence Survey, total score
Exercise perceived capability | 1-year
  Adolescent report on the Physical Activity, Patient-Reported outcome Measurement Information System (PROMIS) Short Form
Depression symptoms | 1-year
  Adolescent report on the 20-item Center for Epidemiologic Studies-Depression Scale (CES-D), total score
Depressive disorder | 1-year
  Schedule for Affective Disorders and Schizophrenia for School-Aged Youth - Computerized Version (KSADS-COMP) interview with adolescent
Eating behavior | 1-year
  Habitual macronutrient/food group intake reported 3 days (2 weekdays, 1 weekend) on the Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA24)
Sleep quality | 1-year
  Adolescent report on the Pittsburgh Sleep Quality Index, total score
Sleep disturbance | 1-year
  Adolescent report on the Insomnia Severity Index, total score
BMI | 1-year
  Derived from height in triplicate by stadiometer and fasting weight by calibrated scale; raw (kg/m2) and z-score/percentile based upon Centers for Disease Control and Prevention (CDC) growth charts
Adiposity | 1-year
  Fat/fat-free mass measured via air displacement plethysmography in a fasted state (BodPod)

OTHER OUTCOMES:
Dispositional mindfulness | 1-year
  Adolescent report on the Mindful Attention Awareness Scale - Adolescent Version (MAAS-A), total score
Weight bias internalization | 1-year
  Adolescent report on the Weight Bias Internalization Scale for Youth (WBIS-Y), total score
Body image | 1-year
  Multidimensional Body Self-Relations Questionnaire Measure composed of 10 subscales: appearance evaluation, fitness evaluation, fitness orientation, health evaluation, health orientation, illness orientation, body areas satisfaction, overweight preoccupation, and self-classified weight.
Automatic thoughts | 1-year
  Adolescent report of frequency of negative and positive thoughts on the Automatic Thoughts Questionnaire (ATQ), negative and positive scale scores
Pleasant activities | 1-year
  Adolescent report on the frequency and perceived pleasantness of physical and social activities on the Pleasant Events Schedule (PES), frequency and pleasantness scales for physical activities and for social activities
Intervention Acceptability | 1-year
  Equal or greater than 80% adolescent liking/credibility ratings (equal or greater than 4 on a scale of 1=not at all to 5=extremely) on a Program Acceptability Questionnaire and themes indicative of liking/perceived benefit on standardized interviews for qualitative coding

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - Colorado State University, Fort Collins, Colorado